CLINICAL TRIAL: NCT00678340
Title: A Single Centre, Randomized, Single Blinded Trial of Wide Area Circumferential Ablation With Pulmonary Vein Isolation Compared to a Multipolar, Circular Ablation Catheter in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Randomized Trial of Two Ablation Catheters in Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pier Lambiase (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); The Royal Bournemouth Hospital (Other)
Responsible Party: Sponsor-Investigator, Pier Lambiase, Chief Investigator, University College London Hospitals
Organization: University College London Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCH 07/0094
Record Dates: First submitted 2008-02-14; First posted 2008-05-15 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Atrial Fibrillation
Keywords: Randomized Controlled Trial; Single-Blind Study; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): WACA and PVI
  Interventions: Device: WACA and PVI
- 2 (Active Comparator): PVAC
  Interventions: Device: PVAC

INTERVENTIONS:
Device: WACA and PVI — Wide area circumferential ablation (WACA) in the pulmonary vein antrum with subsequent pulmonary vein isolation (PVI) with a single tip irrigated catheter.
  Arms: 1
Device: PVAC — Circumferential ablation with a circular ablation catheter (Ablation Frontiers) to electrical silence.
  Other Names: Pulmonary vein ablation catheter, Ablation Frontiers
  Arms: 2

SUMMARY:
Atrial fibrillation (AF) is a chaotic heart rhythm of the top chambers of the heart. AF occurs in up to 10% of the population over the age of 60. It is associated with tiredness, impaired functional capacity and is the cause of up to 10% of strokes.

Ablation is a procedure performed with small tubes (catheters) that are introduced through the top of the leg. Burns are made inside of the heart to treat AF. This procedure has been shown to cure 90% of patients with intermittent (paroxysmal) AF.

The investigators currently use either one of two different catheters to create these burns inside the heart. The investigators do not know which is the best catheter to use in patients with paroxysmal atrial fibrillation.

The investigators study will randomly allocate patients to have their ablation performed by either one of the catheters to give a fair comparison between the two. The investigators objective is to study the differences between these two catheters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal AF with a planned ablation procedure

Exclusion Criteria:

* Prior AF ablation
* LA size greater than 60mm
* Mechanical prosthetic MVR
* Hypertrophic cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2007-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Freedom of AF at 1 year following AF ablation procedure measured by 7 day holter recording | 1 year
Procedural time for pulmonary vein isolation | Index procedure

SECONDARY OUTCOMES:
All procedural complications | Index
Incidence of pulmonary vein stenosis measure by MRI at 6 months post procedure | 6 months
Quality of life questionnaire | 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pier D Lambiase, PhD, Principal Investigator — University College Hospital London NHS Foundation Trust
Locations (1):
- University College Hospital London NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] McCready J, Chow AW, Lowe MD, Segal OR, Ahsan S, de Bono J, Dhaliwal M, Mfuko C, Ng A, Rowland ER, Bradley RJ, Paisey J, Roberts P, Morgan JM, Sandilands A, Yue A, Lambiase PD. Safety and efficacy of multipolar pulmonary vein ablation catheter vs. irrigated radiofrequency ablation for paroxysmal atrial fibrillation: a randomized multicentre trial. Europace. 2014 Aug;16(8):1145-53. doi: 10.1093/europace/euu064. Epub 2014 May 19. PMID 24843051